CLINICAL TRIAL: NCT04001062
Title: Non-operative vs Surgical Treatment of Isolated Non-Thumb Metacarpal Shaft Fractures, A Randomized Controlled Trial
Brief Title: Non-operative vs Surgical Treatment of Isolated Non-Thumb Metacarpal Shaft Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution prior to results being available.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014561
Record Dates: First submitted 2019-06-21; First posted 2019-06-27 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Metacarpal Fracture
Keywords: Metacarpal Shaft Fracture
MeSH Terms: interventions — Surgical Fixation Devices; Fracture Fixation; Conservative Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-operatively (Active Comparator): 1. Adults 18 and older
  2. Native English-speaker
  3. Non-thumb isolated single metacarpal shaft closed fracture (both scissoring and non-scissoring injuries)
  Interventions: Procedure: Surgical Fixation
- Surgical (Active Comparator): 1. Adults 18 and older
  2. Native English-speaker
  3. Non-thumb isolated single metacarpal shaft closed fracture (both scissoring and non-scissoring injuries)
  Interventions: Other: Non-Operative Management

INTERVENTIONS:
Procedure: Surgical Fixation — For both scissoring and non-scissoring injuries surgical fixation by either pinning, dorsal plate, or lag screws will be considered. This will be determined by surgeon expertise at the time of surgical fixation. Postoperative, a volar short arm splint and immediate AROM at full range with buddy taping to adjacent digit will be indicated. Transition to removable short arm splint at week 2 after suture removal. No strengthening until clinical union.
  Other Names: Fracture Fixation
  Arms: Non-operatively
Other: Non-Operative Management — 1. For non-scissoring injuries: Placement of short-arm cast; immediate AROM with buddy taping to adjacent digit. Focus on achieving pulp-to palm distance of <2cm at first visit. Transition to removable short arm splint at week 2 (discontinue at 6 weeks or when non-tender). Strengthening after clinical union.
  2. For scissoring injuries: Closed reduction in clinic/ER and placement of short-arm cast; immediate full range AROM with buddy taping to adjacent digit. Focus on achieving pulp-to palm distance of <2cm at first visit. Transition to removable short arm splint at week 2 (discontinue at 6 weeks or when non-tender). Strengthening after clinical union
  Other Names: Conservative Management
  Arms: Surgical

SUMMARY:
There is a lack of strong evidence guiding the treatment of non-thumb isolated closed metacarpal shaft fractures towards operative fixation versus conservative management. Surgical approach is largely decided by surgeon preference/skill, qualities of fracture, and extent of injury. Previous studies have shown that many metacarpal fractures can be treated non-operatively, with outcomes being as good as or better than those treated with surgery. Surgery using plates can often cause stiffness, contractures, and in rare causes nonunion infection or tendon rupture. This study will seek to build upon previous evidence to help guide future surgeons as they decide how to approach a closed non-thumb metacarpal fractures. Patients will be identified in clinic after x-rays are positive for a non-thumb metacarpal fracture. If they consent to participate in the study, they will be put into either the non-operative or surgical group. This decision will be done through randomization.The investigators anticipate that 100 subjects will be enrolled. Patient reported outcomes, including the PROMIS forms, Disabilities of the Arm, Shoulder and Hand (DASH) surveys and Visual Analog Scale (VAS) will be recorded. Range of motion will be assessed at all time points along with grip strength. X-rays will be evaluated for metacarpal shortening, rotation or non-union. In addition, time for clinical and radiologic union will be documented.

DETAILED DESCRIPTION:
Research Objectives:

The goal of this study is to compare the treatment of outcomes for the nonoperative vs. surgical treatment of isolated closed acute non-thumb metacarpal shaft fracture.

a. Primary Measure: i. Functional outcome: Patient Reported Outcomes, including VAS, PROMIS, DASH (Pre-Op, 2 weeks, 6 weeks, 3 months, 6 months) b. Secondary Measures: i. Grip Strength (6 weeks, 3 months, 6 months) ii. Extensor Lag (degrees) (Pre-Op, 2 weeks, 6 weeks, 3 months, 6 months) iii. Composite range of motion (pulp to palm distance) (Pre-Op, 2 weeks, 6 weeks, 3 months, 6 months) iv. Radiographic metacarpal shortening (at each visit) v. Malrotation (scissoring/gapping) (Pre-Op, 2 weeks, 6 weeks, 3 months, 6 months) vi. Timing of clinical union (lack of tenderness on palpation or stress) vii. Timing of radiographic union (bony bridging across fracture site)

Study Design:

1. Patients will be identified in clinic after x-rays are positive for a non-thumb metacarpal fracture. If they consent to participate in the study, they will be put into either the non-operative or surgical group. This decision will be done through randomization, and the physician will not select which group the patient is in.
2. Pre-operatively, the patient will have the following standard of care procedures:

   1. Patient reported outcomes, including the PROMIS forms and Visual Analog Scale (VAS),
   2. Radiographic measurement of metacarpal shortening
   3. Range of Motion Measurements
   4. Malrotation (scissoring/gapping) measurement
3. Pre-operatively, the patient will have the following procedures as research only:

   a. Disabilities of the Arm, Shoulder and Hand survey (DASH)
4. Surgical Treatment vs. Non-Surgical Treatment Groups

   1. For non-operatively addressed scissoring injuries: Closed reduction in clinic/ER and placement of short-arm cast; immediate full range active range of motion (AROM) with buddy taping to adjacent digit. Focus on achieving pulp-to palm distance of <2cm at first visit. Transition to removable short arm splint at week 2 (discontinue at 6 weeks or when non-tender). Strengthening after clinical union.
   2. For non-operatively addressed non-scissoring injuries: Placement of short-arm cast; immediate active range of motion (AROM) with buddy taping to adjacent digit. Focus on achieving pulp-to palm distance of <2cm at first visit. Transition to removable short arm splint at week 2 (discontinue at 6 weeks or when non-tender). Strengthening after clinical union.
   3. For surgical fixation: The surgeon will utilize either pinning, dorsal plate, or lag screws. This will be determined by surgeon expertise while intra-op. Postoperative volar short arm splint, immediate active range of motion (AROM) at full range with buddy taping to adjacent digit. Transition to removable short arm splint at week 2 after suture removal. No strengthening until clinical union.
5. Post-operatively, the patient will have the following standard of care procedures at the 2 week, 6 week, 3 month and 6 month time points:

   1. Patient reported outcomes, including the PROMIS forms and Visual Analog Scale (VAS)
   2. Radiographic measurement of metacarpal shortening
   3. Range of Motion Measurements
   4. Malrotation (scissoring/gapping) measurement
   5. Grip Strength (at 6 week, 3 month, and 6 month follow-ups only)
   6. Notation of timing of clinical union based upon the lack of tenderness on palpation or stress
   7. Notation of the timing of radiographic union, based on bony bridging across the fracture site
6. Post-operatively, the patient will have the following research only procedures at the 2 week, 6 week, 3 month and 6 month time points:

   a. Disabilities of the Arm, Shoulder and Hand survey (DASH)
7. Treatment failure is defined as non-union. Patients may be removed from the study if they are unable to comply with post-operative requirements, or if their injuries are found to be more complex than the study allows for.
8. If patients are removed from the study prematurely, their treatment will continue as standard of care with their attending physician.

Potential Risks:

A potential risk of this treatment is that a patient will experience a non-union or malunion. This is a normal risk of non-thumb metacarpal fracture.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 and older
* Native English-speaker
* Non-thumb isolated single metacarpal shaft closed fracture

Exclusion Criteria:

* Pre-existing condition in the involved hand/wrist, hand contracture or deformity, pre-existing stiffness
* Cognitive dysfunction with inability to follow rehabilitation protocol
* Subacute/chronic fracture (>4 weeks)
* Pregnant Participants
* VA patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Vas Pain Score | 6 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 being "no pain" and 10 being "worst pain."
PROMIS score | 6 months
  The Patient-Reported Outcomes Measurement Information System® (PROMIS) is a flexible set of tools designed to measure self-reported physical, mental and social health and wellbeing. PROMIS instruments contain a fixed number of items from seven PROMIS domains: depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities. The questionnarie assesses each of the 7 PROMIS domains with 4 questions. The questions are ranked on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity. Norm-based scores are calculated for each domain on the PROMIS measures, so that a score of 50 represents the mean or average of the reference population. A score of 60 means that the person is one standard deviation above the reference population (standard deviation = 10).
Disabilities of the Arm, Shoulder and Hand (DASH) | 6 months
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
Grip Strength | 6 months
  Grip strength will be measured using a Hand Dynamometer with the participants seated, their elbow by their side and flexed to right angles, and a neutral wrist position, the dynamometer handle position II and provision of support underneath the dynamometer. Pressure will be reported in pounds / Kilograms of pressure
Extension lag | 6 months
  Measured with a goniometer and expressed in degrees (°)
Finger Range of Motion | 6 months
  Measured with a goniometer and expressed in degrees (°)
Time to union | 6 months
  Time to achieve clinical and radiologic formation of a stable callus, documented in days
Adverse events | 6 months
  Adverse Events by type over time, severity, seriousness, and relatedness. AEs will be tabulated and summarized as counts and percentages. AEs will also be cross-tabulated according to:
  Severity; Unanticipated Adverse Device Effect (UADE) Seriousness (Serious Adverse Event (SAE), Non-serious AE); Device-Relatedness (Unrelated, Possibly Related, Probably Related, Definitely Related); Procedure-Relatedness (Unrelated, Possibly Related, Probably Related, Definitely Related).

CONTACTS AND LOCATIONS:
Overall Officials: Jay Bridgeman, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No The Investigator will maintain all study records according to applicable University regulatory requirement(s). Hard copy records will be retained for at least 7 years after the last clinic follow-up visit at the Missouri Orthopaedic Institute in a locked filing cabinet. Electronic records will be retained for the same amount of time but on secured computers and servers. If the Investigator withdraws from the responsibility of keeping the study records, custody will be transferred to a person willing to accept the responsibility.

REFERENCES:
- [Background] Macdonald BB, Higgins A, Kean S, Smith C, Lalonde DH. Long-term follow-up of unoperated, nonscissoring spiral metacarpal fractures. Plast Surg (Oakv). 2014 Winter;22(4):254-8. doi: 10.4172/plastic-surgery.1000888. PMID 25535464
- [Background] Eglseder WA Jr, Juliano PJ, Roure R. Fractures of the fourth metacarpal. J Orthop Trauma. 1997 Aug;11(6):441-5. doi: 10.1097/00005131-199708000-00014. PMID 9314153
- [Background] Al-Qattan MM. Outcome of conservative management of spiral/long oblique fractures of the metacarpal shaft of the fingers using a palmar wrist splint and immediate mobilisation of the fingers. J Hand Surg Eur Vol. 2008 Dec;33(6):723-7. doi: 10.1177/1753193408093559. Epub 2008 Jul 28. PMID 18662959
- [Background] Westbrook AP, Davis TR, Armstrong D, Burke FD. The clinical significance of malunion of fractures of the neck and shaft of the little finger metacarpal. J Hand Surg Eur Vol. 2008 Dec;33(6):732-9. doi: 10.1177/1753193408092497. Epub 2008 Oct 20. PMID 18936129
- [Background] Kollitz KM, Hammert WC, Vedder NB, Huang JI. Metacarpal fractures: treatment and complications. Hand (N Y). 2014 Mar;9(1):16-23. doi: 10.1007/s11552-013-9562-1. PMID 24570632
- [Result] Giddins GE. The non-operative management of hand fractures. J Hand Surg Eur Vol. 2015 Jan;40(1):33-41. doi: 10.1177/1753193414548170. Epub 2014 Sep 12. PMID 25217094
- [Result] Khan A, Giddins G. The outcome of conservative treatment of spiral metacarpal fractures and the role of the deep transverse metacarpal ligaments in stabilizing these injuries. J Hand Surg Eur Vol. 2015 Jan;40(1):59-62. doi: 10.1177/1753193414540408. Epub 2014 Jun 23. PMID 24963083